CLINICAL TRIAL: NCT01835314
Title: Compassionate Use of Stiripentol in Dravet Syndrome
Status: No longer available | Type: Expanded Access
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0315
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — stiripentol

INTERVENTIONS:
Drug: Stiripentol — Stiripentol 5-50mg/kg/d divided twice or three times a day by mouth

SUMMARY:
Compassionate use of Stiripentol in Dravet Syndrome. This is a treatment protocol, not a research study, therefore children will only be monitored on a clinical basis for seizure improvement predominantly by parent and caregiver report.

DETAILED DESCRIPTION:
This is a treatment protocol for compassionate use, not a research study, therefore children will only be monitored on a clinical basis for seizure improvement predominantly by parent and caregiver report.

ELIGIBILITY:
Children with genetic confirmation of Dravet syndrome (a documented sodium channel, voltage-gated, type I, alpha subunit (SCN1A) mutation) or clinical confirmation of Dravet syndrome by two pediatric neurologist will be considered to have Dravet syndrome. In order to enter the treatment protocol there will be documented treatment failure of at least two therapeutic anticonvulsants excluding Na channel blockers. Anticonvulsants that are Na channel blockers such as carbamazepine and lamotrigine as known to provoke seizures in this patient population.

Ages: 1 Year to 21 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Knupp, MD, Principal Investigator — University of Colorado/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States